CLINICAL TRIAL: NCT06181734
Title: Ivosidenib in Combination With Azacitidine as First-line Treatment for Adult Patients With Newly Diagnosed AML With an IDH1 R132 Mutation Who Are Not Eligible to Receive Standard Induction Chemotherapy
Brief Title: Ivosidenib (TIBSOVO®) Combined With Azacitidine According to Current SmPC
Acronym: CONFIDHENCE
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: iOM-070496
Record Dates: First submitted 2023-11-27; First posted 2023-12-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: IDH1 R132 mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ivosidenib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ivosidenib — inhibitor of mutant IDH1

SUMMARY:
The goal of this non-interventional study is to evaluate quality of life (QoL) in adult patients with newly diagnosed IDH1 R132-mutated AML who are not eligible to receive standard induction chemotherapy and who are treated with ivosidenib in combination with azacitidine in a real-world setting in Germany.

The main questions it aims to answer are:

* Evaluate QoL by validated and widely used Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) questionnaire and European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) questionnaire during treatment and follow-up period
* Assesment of effectiveness in routine treatment (e.g. overall survival, event-free survival, overall response rate)
* Assessment of drug safety (all adverse events)
* Description of treatment reality in detail

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Newly diagnosed Acute Myeloid Leukemia (AML).
* Having an isocitrate dehydrogenase 1 (IDH1) R132 mutation.
* Not eligible to receive standard induction chemotherapy.
* Decision for treatment with ivosidenib in combination with azacitidine as per current SmPC.
* Signed written informed consent*

  *Patients are allowed to be enrolled up to 6 weeks after ivosidenib plus azacitidine dose
* For patients participating in PROs: Willingness and capability to participate in PRO assessment in German language
* Other criteria according to current SmPC.

Exclusion Criteria:

* Participation in an interventional clinical trial within 30 days prior to enrollment or simultaneous participation in an interventional clinical trial except for the follow-up period.
* Patients unable to consent
* Other contraindications according to current SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with newly diagnosed, IDH1 R132- mutated AML who are not eligible to receive standard induction chemotherapy and with treatment decision for ivosidenib in combination with azacitidine according to SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Evaluate quality of life | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Validation of FACT-Leu. Change from baseline (treatment start) of FACT-Leu total score over time

SECONDARY OUTCOMES:
Subjective well-being: Validation of FACT-Leu | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Change from baseline (treatment start) of FACT-Leu subscale score over time
Subjective well-being: Validation of FACT-Leu | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Change from baseline (treatment start) of FACT-G total scores over time
Subjective well-being: Validation of FACT-Leu | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Change from baseline (treatment start) of Trial outcome Index over time
Subjective well-being: Validation of FACT-Leu | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Time to deterioration of FACT-Leu total score
Subjective well-being: Validation of FACT-Leu | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Time to deterioration of FACT-G total score
Subjective well-being: Validation of FACT-Leu | Baseline until end of study (during ivosidinib treatment and Follow-Up); Up to 54 months
  Time to deterioration of Trial Outcome Index
Subjective well-being: Validation of FACT-Leu and EQ-5D-5L questionnaire | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  FACT-Leu total score over time over time
Subjective well-being: Validation of FACT-Leu and EQ-5D-5L questionnaire | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  FACT-G total score over time
Subjective well-being: Validation of FACT-Leu and EQ-5D-5L questionnaire | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Trial Outcome Index
Subjective well-being: Validation of EQ-5D-5L questionnaire | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Change from baseline of the EQ-5D-5L visual analogue scale score over time
Subjective well-being: Validation of EQ-5D-5L questionnaire | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  EQ-5D-5L visual analogue scale score over time
Subjective well-being: Validation of EQ-5D-5L questionnaire | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Index value of EQ-5D-5L over time
Subjective well-being: Validation of EQ-5D-5L questionnaire | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Time to deterioration of the EQ-%D-5l visual analogue scale score over time
Assesment of effectiveness in routine treatment | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Assesment of overall survival (OS),
Assesment of effectiveness in routine treatment | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Event-free survival (EFS)
Assesment of effectiveness in routine treatment | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Overall Response Rate (ORR; i.e. CR, CR with incomplete hematologic recovery (Cri), (including CR with incomplete platelet recovery (CRp), CR with partial hematologic recovery (CRh), or partial recovery (PR)), Duration of CR (DOCR), Duration of Response (DOR; CR, Cri, CRp, CRh, PR))
Assesment of effectiveness in routine treatment | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Time to first response (TTR)
Assessment of drug safety | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Assesment of adverse events (AEs), serious adverse events (SAEs), adverse drug reactions (ADRs), serious adverse drug reactions (SADRs), Adverse events of special interest (AESIs)
Assessment of parameters of treatment decision making | From date of patient enrollment until start of treatment
  Frequency of distinct parameters affecting therapy choice including reasons why patient is ineligible for standard induction chemotherapy.
Ivosidenib and azacitidine treatment: Dose intensity | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Descriptive statistics will be provided for dose intensity for ivosidinib and azacitidine
Ivosidenib and azacitidine treatment: Frequency and type of dose modification | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Frequency tables will be provided for frequency and type of dose modification for ivosidinib and azacitidine
Ivosidenib and azacitidine treatment: Reason for dose modifications | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Frequency tables of reasons for dose modifications will be provided for ivosidinib and azacitidine
Ivosidenib and azacitidine treatment: Duration of treatment in total and for each substance | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Descriptive statistics will be provided for duration of treatment in total and for each substance dose
Ivosidenib and azacitidine treatment: Reason for end of treatment (EOT) | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Frequency tables of EOT-reasons will be provided
Treatment reality in detail: Transfusion dependency | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Proportion of transfusion dependent patients to independency and vice versa will be provided
Treatment reality in detail: Concomitant medication | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Frequency table of concomitant medication in total and frequency of concomitant medications known to induce QT prolongation (e.g., antiarrhythmic medicines, fluoroquinolones, triazole anti-fungals, 5-HT3 receptor antagonists) as well as strong CYP3A4 inducers or dabigatran will be provided
Treatment reality in detail: Subsequent antineoplastic therapies | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Description of frequency and type of subsequent antineoplastic therapies by line of therapy (number and substance)
Treatment reality in detail: Frequency of hospitalizations/emergency room visits | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Frequency table of hospitalization and emergency room visits will be provided
Treatment reality in detail: Reasons for hospitalizations/emergency room visits | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Frequency table of reasons for hospitalization and emergency room visits will be provided
Treatment reality in detail: Length of hospital stay | Baseline until end of study (during ivosidenib treatment and Follow-Up); Up to 54 months
  Descriptive statistic for length of hospital stay will be provided

CONTACTS AND LOCATIONS:
Locations (1):
- Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No